CLINICAL TRIAL: NCT04552548
Title: Ultrasound-Guided Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Analgesia in Children Undergoing Laparoscopic Surgery.
Brief Title: Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Analgesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, haidy salah mansour, Professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 271:7/2019
Record Dates: First submitted 2020-08-31; First posted 2020-09-17 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): the patients will receive regular analgesics (1 µg /kg fentanyl with induction and 15mg/kg paracetamol before extubation)
- TAP group (Active Comparator): the patients will receive bilateral TAP block using (0.5 ml/ kg bupivacaine 0.25%) in each side + regular analgesics.
  Interventions: Other: regional nerve block
- quadratus lumborum group (Active Comparator): the patients will receive bilateral quadratus lumborum block using (0.5 ml/ kg bupivacaine 0.25%) in each side + regular analgesics.
  Interventions: Other: regional nerve block

INTERVENTIONS:
Other: regional nerve block — Abdominal field blocks have been used in anesthesia for surgery involving the anterior abdominal wall with ultrasound-guided technique. TAP block is a regional anesthetic technique that blocks neural afferents of the anterolateral abdominal wall. Using anatomical landmark guidance or with the aid of ultrasound (US), local anesthetic is injected into the transversus abdominis fascial plane, where the nerves from T6 to L1 are located. Ultrasound-guided quadratus lumborum (QL) block is considered now as one of the novel truncal abdominal blocks, as it is effective in preventing somatic pain associated with upper and lower abdominal surgeries.
  Arms: TAP group; quadratus lumborum group

SUMMARY:
The aim of the present study is to evaluate and compare the analgesic effect of ultrasound-guided Quadratus Lumborum Block with ultrasound-guided Transversus Abdominis plane block in pediatric Laparoscopic lower abdominal surgeries

DETAILED DESCRIPTION:
90 male and female patients aged from 1 to 7 years old from ASA class I to II undergoing elective laparoscopic lower abdominal surgery will be randomly divided into three equal groups of thirty patients each by using computer generated random table.

Technique of the study After insertion of venous access, all children received premedication in the form of atropine at a dose of 0.01-0.02 mg/kg. Perioperative monitoring included continuous ECG, pulse oximetry and non-invasive arterial blood pressure. Baseline reading of heart rate, mean arterial blood pressure was recorded after monitor attachment. General anesthesia will be induced using propofol 1.5-2.5 mg/kg over 20-30 sec. as tolerated, atracurium 0.5 mg/kg to facilitate endotracheal intubation and fentanyl 1 µg/kg. Anesthesia will be maintained using isoflurane (1 MAC) and atracurium 0.1 mg/kg supplements will be given to maintain muscle relaxation.

TAP block or quadratus lumborum block will be performed in all patients immediately after induction and before starting of surgery. patients will be allocated randomly into three equal groups , 30 patients in each as the following :-

Group C "Control group" will receive regular analgesics (1 µg /kg fentanyl with induction and 15mg/kg paracetamol before extubation).

Group TAP "TAP group" will receive bilateral TAP block using (0.5 ml/ kg bupivacaine 0.25%) in each side + regular analgesics.

Group QL"quadratus lumborum group" will receive bilateral quadratus lumborum block using (0.5 ml/ kg bupivacaine 0.25%) in each side + regular analgesics.

TAP block procedure

With the patient in the supine position, the site of the ultrasound and needle entry was sterilized. The TAP block will be performed laterally behind the midaxillary line between the iliac crest and the most inferior extent of the ribs. The plane between the internal oblique and transversus abdominis muscle located around the midaxillary line with the probe transverse to the abdomen. Anteriorly, the needle passes to come perpendicular to the ultrasound beam and placed between transversus and internal oblique posterior to the midaxillary line. Then, the local anesthetic will be injected. QL block prcedure

bilateral ultrasound guided transmuscular quadrates lumborum (TQL) block was given SONOSITE NANOMAX; the scanning probe was the linear 25N multifrequency 13-6 MHz transducer (L25x13-6 MHz linear array) made in USA. In lateral position, the side to be blocked was kept up and probe was placed in the midaxillary line in the transverse plane immediately above the iliac crest and then it was slided dorsally till the Shamrock sign was clearly identified. In "Shamrock sign" The quadratus lumborum (QL) muscle is seen as a superior leaf of the Shamrock at the apex of the transverse process (TP) of L4, erector spinae (ES) muscles make up the posterior leaf, psoas major (PM) muscle makes the anterior leaf and the transverse process (TP) represents the stem connecting the 3leaves. A 22-G 90-mm spinal needle was inserted from the posterior end of the probe and directed for the fascial plane between the QL and PM muscles through the QL muscle. Once needle was confirmed at correct location the drug was injected. Other side was also injected in similar manner. The parents were not aware of group allocation as the block was done after induction of anesthesia. An independent anesthesiologist conducted postoperative assessments and was not aware of group allocation

The surgical intervention was started 15 min after QL block. Pneumoperitoneum was maintained at a flow rate of 0.5 L/min and a pressure of 8-12 mm Hg with CO2 insufflation.

After completion of surgical procedure anesthesia was discontinued, muscle relaxant reversed using atropine 0.02 mg/kg and 0.05 mg/kg of prostigmine. Paracetamol infusion (15 mg/kg) will be given by intravenous infusion before extubation. After extubation transfer the children to PACU.

Postoperatively pain will be assessed using FLACC score (face, leg, activity, cry and consolability) as shown in the table below. Acetaminophine (perfalgan) 15 mg/kg IV will be given as rescue analgesia for patients if FLACC score >4.

Parameters will be assessed

A. Preoperative and intraoperative measurements:

1. Hemodynamic parameters: HR, MAP and SaO2 were recorded before and immediately after induction of anesthesia, at the time of puncture of the prop and then every 5 min intervals until the end of the operation.
2. Analgesic requirement: all through the procedure (by measuring the analgesic need intra operative in the form of fentanyl 0.5 µg/kg) in case of increase in intraoperative mean arterial blood pressure or heart rate of more than 20% of baseline for longer than 5 minutes.
3. Incidence of complications: in the form of hemodynamic instability, injury to the underlying structures, and hematoma formation as recorded under ultrasound guidance.

B. Postoperative measurement:

1. The number of patients who require rescue analgesia in the first 24 h. 2. Quality of analgesia: it will be assessed immediately postoperatively, every 30min in the PACU and then at 4, 6, 8, 10, 12, 18, and 24 h postoperatively using FLACC score.

3. Time to the first analgesic requirement: Duration of analgesia was defined as the time interval from completion of local anesthetic administration till first need of rescue analgesic (FLACC>4) in the form of IV paracetamol 15mg/kg.

Each category is scored on the 0-2 scale, which results in a total score of 0-10. 0 Relaxed and comfortable 1-3 Mild discomfort Behaviour 0 1 2 Face No particular expression or smile

Occasional grimace or frown, withdrawn, disinterested

Frequent to constant quivering chin, clenched jow Legs Normal position or relaxed

Uneasy, restless, tense Kicking or legs drawn up Activity Lying quietly, normal position, moves easily

Squirming, shifting, back and forth, tense

Arched, rigid or jerking Cry No cry (awake or asleep)

Moans or whimpers; occasional complaint

Crying steadily, screams, sobs, frequent complaints Consolability Content, relaxed Reassured by touching, hugging or being talked to, distractible Difficult to console or comfort 4-6 Moderate pain 7-10 Severe discomfort or pain or both (Merkel, et al., 1997) 4. Total amount and the numbers of analgesic doses in 24h. 5. Hemodynamic data: HR, MAP and SaO2 were recorded up to 120 min.

6. length of hospital stay and patients or parents satisfaction assessed on a 5point scale. 1-completely dissatisfied, 2-dissatisfied, 3-not satisfied nor dissatisfied, 4- satisfied 5-completely satisfied 7. Postoperative complication: including postoperative hypotention or bradycardia (decrease in MAP or HR by more than 20% of baseline value), postoperative nausea and vomiting (PONV).

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II physical status patients
* Children scheduled for laparoscopic surgery
* Duration of Laparoscopic procedure not exceeding 90 minutes

Exclusion Criteria:

* Sensitivities to local anesthetics
* Significant renal, liver, or cardiac disease
* Surgery requiring an open procedure
* Participants refusing regional block
* Those having bleeding disorders, skin lesions or wounds at the site of proposed needle insertion, evidence of peritonitis, septicemia
* Children required emergency procedures.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
quality of postoperative analgesia | 24 hours after surgery
  Postoperative Pain scores as FLACC score (face, legs, activity, cry and consolability)

SECONDARY OUTCOMES:
analgesic consumption | 24 hours
  Total postoperative analgesic consumption : The total paracetamol (mg/kg)
duration of analgesia | 24 hours after block
  Time to first demand of rescue analgesic: Duration of analgesia was defined as the time interval from completion of local anesthetic administration till first need of rescue analgesic (FLACC>4) in the form of IV paracetamol 15mg/kg.

CONTACTS AND LOCATIONS:
Locations (1):
- Minya University, Minya, Egypt